CLINICAL TRIAL: NCT05766995
Title: Efficacy of Three Oral Self-care Regimens on Clinical Parameters of Inflammation and Plaque: Part 1 - a Four Week Randomized Controlled Trial
Brief Title: Evaluation of 3 Oral Self-care Regimens on Clinical Signs of Inflammation and Plaque
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Water Pik, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2021-WP-1
Record Dates: First submitted 2023-01-09; First posted 2023-03-13 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-01

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Manual toothbrush and water flosser with standard jet tip (Experimental): Brush with a standard ADA manual toothbrush twice daily followed by water flossing once in the evening
  Interventions: Device: Waterpik Water Flosser
- Manual toothbrush and water flosser with targeted jet tip (Experimental): Brush with a standard ADA manual toothbrush twice daily followed by water flossing once in the evening
  Interventions: Device: Oral-B Water Flosser
- Manual toothbrush and dental floss (Active Comparator): Brush with a standard ADA manual toothbrush twice daily followed by dental flossing once in the evening
  Interventions: Device: Waxed Dental Floss

INTERVENTIONS:
Device: Waterpik Water Flosser — A pulsating water flosser and jet tip designed to clean between the teeth and below the gingival margin.
  Other Names: dental water jet; oral irrigator
  Arms: Manual toothbrush and water flosser with standard jet tip
Device: Oral-B Water Flosser — A water flosser and specialized tip that delivers water with microbubbles of air
  Other Names: dental water jet; oral irrigator
  Arms: Manual toothbrush and water flosser with targeted jet tip
Device: Waxed Dental Floss — Nylon string used to clean between the teeth manually
  Arms: Manual toothbrush and dental floss

SUMMARY:
To compare three different oral hygiene regimens on changes in gum tissue appearance, gum bleeding, and plaque scores.

DETAILED DESCRIPTION:
The goal of this clinical trial was to compare the effect of different battery powered water in and adult population with mild to moderate gingivitis. The main questions it aims to answer are:

* Is there a difference between the two water flosser devices on gum bleeding scores?
* Is there a difference between the two water flosser devices on plaque accumulation and removal?
* Is there a difference between the two water flosser devices on signs of gingivitis?

Researchers will compare the two groups using a water flosser (experimental) to see how it compares to traditional brushing and flossing (control).

ELIGIBILITY:
Inclusion Criteria:

* Have provided written informed consent prior to being entered into the study.
* Be between 18 and 75 years of age, male or female.
* Have at least twenty (20) natural teeth (5 evaluable in each quadrant) with scorable facial and lingual surfaces as determined by the clinical examiner.
* Nonsmoking (assessed as < 1 cigarette every day for at least a year).
* Have a mean baseline plaque index score of ≥0.60 as determined by the Rustogi Modification of the Navy Plaque Index (RMNPI).
* Have a mean baseline gingival index score of ≥1.75 as determined by the Modified Gingival Index (MGI).
* Have a mean bleeding on probing score of 50%.
* Have probe readings ≤4 mm.
* Agree not to have a dental prophylaxis or any other elective, non-emergency dental procedures any time during the study.
* Agree to abstain from the use of chewing gum, mouth rinses, any toothpaste other than the study toothpaste, tooth whitening products (either professional or at home use) and all other oral hygiene other than the study procedures for the duration of the study.
* Agree to refrain from all oral hygiene on the morning of each evaluation visit and to refrain from eating, drinking or chewing gum for 4 hours prior to each evaluation visit.
* Agree to comply with the conditions and schedule of the study.

Exclusion Criteria:

* Physical limitations or restrictions that might preclude normal use of devices.
* Evidence of gross oral pathology, including widespread caries or chronic neglect, extensive restoration, pre-existing gross plaque or soft or hard tissue tumor of the oral cavity.
* Supra- or subgingival calculus that might interfere with evaluations as determined by the clinical examiner.
* Evidence of major oral hard or soft tissue lesions or trauma at the baseline visit as determined by the clinical examiner.
* Conditions requiring antibiotic treatment prior to dental procedures.
* History of uncontrolled diabetes or hepatic or renal disease, or other serious conditions or transmittable disease, (e.g. COVID-19, AIDS).
* Subjects with grossly carious, fully crowned, or extensively restored teeth, orthodontic appliances, peri/oral piercings, or removable partial dentures.
* Treatment with antibiotics within the 1-month period before the baseline examination, or a condition that is likely to require antibiotic treatment over the course of the trial.
* Chronic treatment (2-weeks or more) with any medication known to affect periodontal status (including phenytoin, calcium antagonists, cyclosporine, Coumadin, nonsteroidal anti-inflammatory drugs, and aspirin (325 mg)) within 1- month of the baseline examination. All other medications for chronic medical conditions must have been initiated at least 3 months before enrollment.
* Have moderate to severe periodontal disease or being actively treated for periodontal disease.
* Concomitant periodontal therapy other than prophylaxis in the last 6 months.
* Professional prophylaxis within 1 month prior to the baseline clinical evaluation.
* Subjects who participate in a gingivitis study in the past month.
* History of significant adverse event following use of oral hygiene products such as toothpastes and mouth rinses.
* Subjects who are allergic to any ingredients in Crest® Cavity Protection or Colgate® Cavity Protection toothpaste.
* Self-reported pregnancy or lactating women since hormonal changes can exaggerate gingival response to dental plaque.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2021-08-03 (Actual); Primary Completion 2021-09-03 (Actual); Study Completion 2021-09-03 (Actual)

PRIMARY OUTCOMES:
Bleeding on probing | 4 weeks
  Bleeding recorded on 6 sites per tooth within 30 seconds of instrumentation. 0 = no bleeding, 1= bleeding. Bleeding determined by number of sites bleeding divided by total number of sites = percent bleeding

SECONDARY OUTCOMES:
Modified gingival index | 4 weeks
  Visual assessment of the gingival tissue. 0 = absence of inflammation, 1 = mild inflammation (slight change in color, little change in texture of any porting of but not the entire marginal or papillary gingival area), 3 = moderate inflammation (glazing, redness, edema, and/or hypertrophy of the marginal or papillary gingival area), 4 = severe inflammation (marked redness, edema and/or hypertrophy of the marginal or papillary gingival area, spontaneous bleeding, congestion, or ulceration.
Rustogi Modification of Navy Plaque Index | 4 weeks
  Plaque is assessed for each tooth area (divided into 9 sections labeled A through I) and scored using the following scale: 0 = absent, and 1 = present. Facial and lingual surfaces of all gradable teeth are scored and a mean plaque index is calculated for each subject at each examination. Subjects' scores were calculated for whole mouth (A through I), along the gingival margin (A through C), and at the proximal (approximal) areas (D and F).

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Mancinelli Lyle, Principal Investigator — Water Pik, Inc.
Locations (1):
- All Sum Research Center Ltd., Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No